CLINICAL TRIAL: NCT07029516
Title: A Randomized, Double Blind, Placebo-controlled, Unicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of a Multi-funtion Toe Nail Patch in Patients Affected by Nail Fragility, Nail Mychosis and Psoriasis
Brief Title: Study to Assess Efficacy, Safety and Tolerability of a Nail Patch in Patients With Nail Fragility, Mychosis, Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wooshin Labottach Co., Ltd. (Industry)
Collaborators: Nextrasearch S.r.l.s. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/AFCV/WOOSHIN/MFP/PL
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Nail Psoriasis; Nail Damage; Mycosis
Keywords: ONICOMYCOSIS; PATCH; UREA; PSORIASIS
MeSH Terms: conditions — Mycoses; Psoriasis

STUDY DESIGN:
Intervention Model Description: 6 GROUPS (3 PATOLOGIES ONE EXPERIMENTAL, ONE PLACEBO)
Who Masked: Participant
Masking Description: ANONIMIZATION
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL COSMETIC (Experimental): APPLICATION OF THE EXPERIMENTAL PATCH WITH COSMETIC
  Interventions: Other: Cosmetic patch containing urea applicated daily for 3 months
- Placebo (Placebo Comparator): Application of the Placebo patch
  Interventions: Other: Placebo patch application

INTERVENTIONS:
Other: Cosmetic patch containing urea applicated daily for 3 months — Daily application of the patch on toes, 3 months treatment
  Arms: EXPERIMENTAL COSMETIC
Other: Placebo patch application — Daily application of a placebo patch on toes for a 3 months treatment
  Arms: Placebo

SUMMARY:
A randomized, double blind, placebo-controlled, unicenter, parallel group study to assess the efficacy, safety and tolerability of a multi-funtion toe nail patch in patients affected by nail fragility, nail mychosis and psoriasis 72 patients in 6 subgroups Treatment duration 3 months + 1 month follow-up

DETAILED DESCRIPTION:
A randomized, double blind, placebo-controlled, mono center, parallel group study.

72 Eligible patients will receive Hydrogel Nail Patch every day for three months, in the evening. All the patients will be characterized according to the percentage of target nail involvement (defined as either 50% or 51-75).

Patients applied their allocated treatment to the surface of all affected nails, in particular Hydrogel Nail Patch or Placebo will be applied topically in the evening at bedtime and taken away in the morning, every day for 12 (twelve)weeks. The subjects will receive a visit by the Clinical Investigator after 4 weeks from the end of treatments.

A single affected nail with Fragility nail or onychomycosis or nail psoriasis will be identified as the target nail for all assessments. Target nails had to fulfil the study's inclusion and exclusion criteria and the presence of nail pathology confirmed by Score Index test, photographic documentation, physician judgement. Patients will attend visits at screening(V0), baseline (V1), and at weeks 3(V2), 6(V3), 9(V4) and 12(V5).

The Multi-Function Toe Nail Patch and the Placebo will be applied topically on the big toe affected by nail pathology, according to their characteristics.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older Fragility Nails Distal Subungual Onychomycosis Nail Psoriasis affecting ≤75% of the nail bed according to a photographic documentation and to a subjective evaluation by the Investigator.

Exclusion Criteria:

* Patients that have proximal subungual onychomycosis, if their distal subungual onychomycosis is extended into the proximal portion of the nail or if it affects >75% of the nail.
* Patients with conditions known to cause abnormal nail appearance, immunosuppression and signs of severe peripheral circulatory insufficiency
* Patients who had used topical antifungal, anti-psoriasis nail treatment within one month or systemic antifungal treatment within three months.
* Patients who have participated in another clinical nail study during the previous three months
* Patients who have a known allergy to any of the study treatments.
* Patients with unrelated nail disorders: onychomycosis, nail psoriasis, genetically induced onychodystrophy.
* Patients with other nail disorders, active or severe psoriasis elsewhere, other autoimmune or inflammatory diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation, based on adverse events numeber of the Multi-Function Hydrogel Nail Patch safety in adult humans affected by Fragility Nails, Onychomycosis and Nail Psoriasis | From the enrollment day (visit 1) to the follow-up visit after 4 months
  Checking of any adverse event during the treatment, and at monthly visits

SECONDARY OUTCOMES:
Efficacy of the patch, measuring the size of the nail patology | From enrollment day (visit 1) to the follow-up visit after 4 months
  Evaluation of the Multi-Function Hydrogel Nail Patch medical device in adult humans affected by Fragility Nails, Onychomycosis and Nail Psoriasis Visual improvement in clear nail at least of 50% considering the number of patients with 50% nail clearing and the rate at which the nail clearing takes place in the two treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Dermatologica - Policlinico - Università degli Studi di Milano Via Francesco Sforza- Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol, CSR
Time Frame: after the publication nontime limit
Access Criteria: TBDefined